CLINICAL TRIAL: NCT03784391
Title: Effectiveness of Nifurtimox in Patients With Chagas' Disease Based on Data From Patient Medical Records in Argentina: a Retrospective Medical Chart Review Study
Brief Title: Study on Benefits of Therapy With Nifurtimox in Chagas Disease, a Parasitic Illness Mostly Transmitted to Humans by a Bug, Using Information From Patient Medical Records in Argentina
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20302
Record Dates: First submitted 2018-12-20; First posted 2018-12-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Chagas' Disease
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment: Patients diagnosed with acute and chronic Chagas' disease, respectively, who were treated with nifurtimox
  Interventions: Drug: Lampit (Nifurtimox, BAYA2502)
- Reference: Patients diagnosed with acute and chronic Chagas' disease, respectively, who did not receive antitrypanosomal treatment

INTERVENTIONS:
Drug: Lampit (Nifurtimox, BAYA2502) — Nifurtimox is a drug already approved in some South American countries since more than 45 years
  Groups: Treatment

SUMMARY:
The researchers in this trial want to analyze prerecorded patient data which provide information on benefits of the drug nifurtimox in patients with a sudden (acute) and long lasting (chronic) Chagas´ disease an illness caused by parasites mostly transmitted to humans by a bug. They also want to learn how often organs, especially the heart, are affected by the illness in treated and untreated chronic Chaga's patients. In order to find this out medical records of adult and pediatric patients in Argentina will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥0 years at time of diagnosis with Chagas' disease
* Diagnosis of Chagas' disease confirmed by parasitological and/or serological method(s) before start of antitrypanosomal treatment or during the course of this antitrypanosomal treatment cycle for the first episode recorded.

Exclusion Criteria:

* Treatment with antitrypanosomal agent(s) other than nifurtimox, including experimental investigational products for Chagas' disease or antitrypanosomal combination treatment
* Patients with known evidence of organ manifestation of chronic Chagas' disease, e.g.Chagas' disease-related cardiomyopathy/heart disease, Chagas' disease-related digestive disease at time of primary diagnosis.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise adult and pediatric patients diagnosed with Chagas' disease, respectively, who were treated with nifurtimox (nifurtimox groups). An untreated reference group comprising adult patients diagnosed with chronic Chagas' disease, who did not receive antitrypanosomal treatment will be considered.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Parasitological cure of adult patients with chronic Chagas' disease | Retrospective analysis from late 1960s to about 1980
  Change in the laboratory test result for Chagas' disease to negative after treatment with nifurtimox and without antitrypanosomal treatment compared to baseline.
  Adults are defined as patients who were 18 years or older at the time of initial diagnosis of acute or chronic Chagas' disease

SECONDARY OUTCOMES:
Parasitological cure of pediatric patients with acute and chronic Chagas' disease | Retrospective analysis from late 1960s to about 1980
  Change in the laboratory test result for Chagas' disease to negative after treatment with nifurtimox and without antitrypanosomal treatment compared to baseline.
  Pediatric population will comprise patients aged 0 to below 18 years at the time of initial diagnosis of acute or chronic Chagas' disease
Occurrence of cardiac manifestations in patients with chronic Chagas' disease | Retrospective analysis from late 1960s to about 1980
  Change from a lower to a more advanced Kuschnir group or cardiac death (change of clinical group) and appearance of new abnormalities on ECG compared to baseline.
Treatment of Cardiomyopathy and/or Heart Failure | Retrospective analysis from late 1960s to about 1980

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Argentina

REFERENCES:
- [Derived] Vizcaya D, Grossmann U, Kleinjung F, Zhang R, Suzart-Woischnik K, Seu S, Ramirez T, Colmegna L, Ledesma O. Serological response to nifurtimox in adult patients with chronic Chagas disease: An observational comparative study in Argentina. PLoS Negl Trop Dis. 2021 Oct 4;15(10):e0009801. doi: 10.1371/journal.pntd.0009801. eCollection 2021 Oct. PMID 34606501
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com